CLINICAL TRIAL: NCT02399696
Title: Primary Care-Based Mindfulness Intervention for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse VA Medical Center (U.S. Federal Agency)
Collaborators: Syracuse University (Other)
Responsible Party: Principal Investigator, Kyle Possemato, Clinical Research Psychologists, Syracuse VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 540
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care-Brief Mindfulness Program (Experimental): A 4-week group program adapted from the 8-week Mindfulness Based Stress Reduction (MBSR) curriculum.
  Interventions: Behavioral: Primary Care-Brief Mindfulness Program
- Primary Care-Treatment as Usual (Active Comparator): Typical VA primary care treatment, including mental health services delivered by primary care staff.
  Interventions: Behavioral: Primary Care-Treatment as Usual

INTERVENTIONS:
Behavioral: Primary Care-Brief Mindfulness Program — A 4-week group program adapted from the 8-week Mindfulness Based Stress Reduction (MBSR) curriculum
  Arms: Primary Care-Brief Mindfulness Program
Behavioral: Primary Care-Treatment as Usual — Typical VA primary care treatment, including mental health services delivered by primary care staff.
  Arms: Primary Care-Treatment as Usual

SUMMARY:
Primary care patients typically do not receive adequate PTSD treatment because of their reluctance to engage in empirically-supported treatments offered in specialty care settings. Effective treatments for PTSD are also typically not provided in primary care. Brief skill-based treatments offered in primary care may alleviate symptoms and prepare patients to engage in additional treatment. VA primary care patients with PTSD (N=62) were recruited for a randomized clinical trial comparing a Primary Care-Brief Mindfulness Program (PC-bMP) to primary care-treatment as usual (PC-TAU). PC-bMP is a 4-week group program adapted from the 8-week Mindfulness Based Stress Reduction (MBSR) curriculum. Veterans in the PC-bMP condition demonstrated significantly greater decreases in PTSD and depressive symptoms from pre-treatment to post-treatment compared to PC-TAU. These gains were maintained at 8 and 12 week follow-up. PC-bMP participants experienced clinically significant decreases in PTSD, averaging a 15-point drop on the Clinician-Administered PTSD Scale. Exploratory analyses revealed that the describing, non-judging, and acting with awareness facets of mindfulness may account for decreases in PTSD. Our data support preliminary efficacy of a brief mindfulness-based intervention for Veterans with PTSD in primary care. Further research is needed to investigate how PC-bMP may facilitate engagement into full length empirically-supported treatment for PTSD.

ELIGIBILITY:
Inclusion Criteria:

1) sub-threshold or diagnostic level PTSD related to military service as determined by the Clinician Administered PTSD Scale

Exclusion Criteria:

1) gross cognitive impairment, 2) moderate to severe traumatic brain injury, 3) suicide attempt or intent to commit suicide in the last two months, and 4) receipt of mental healthcare (psychotherapy or medication) outside VA primary in the last two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms as measured by the PTSD Checklist | 8 weeks

SECONDARY OUTCOMES:
Depression symptoms as measured by the Patient Health Questionaire-9 | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Possemato, Ph.D., Principal Investigator — Syracuse VAMC